CLINICAL TRIAL: NCT01682538
Title: A Study to Evaluate the Bioequivalence of Orfadin Suspension 4 mg/mL Compared to Orfadin Capsules 10 mg, and the Effect of Food on the Bioavailability of the Suspension. An Open-label, Randomized, Cross-over, Single-dose Study in Healthy Volunteers
Brief Title: Bioequivalence of Orfadin Suspension Compared to Orfadin Capsules, and the Effect of Food on the Bioavailability of the Suspension
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Swedish Orphan Biovitrum (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Sobi.NTBC-001
Record Dates: First submitted 2012-09-07; First posted 2012-09-11 (Estimated); Results first posted 2014-02-20 (Estimated); Last update posted 2014-03-17 (Estimated); Status verified 2014-02

CONDITIONS: Healthy Volunteers
Keywords: Orfadin; Nitisinone; Bioequivalence; Bioavailability
MeSH Terms: interventions — nitisinone; Capsules; Suspensions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Orfadin capsules, fasting (Active Comparator): Orfadin capsules, single dose, 30 mg
  Interventions: Drug: Nitisinone, capsule
- Orfadin suspension, fasting (Experimental): Orfadin suspension 4 mg/mL, single dose 30 mg (7,5 mL)
  Interventions: Drug: Nitisinone, suspension
- Orfadin suspension, with food (Experimental): Orfadin suspension 4mg/mL, single dose 30 mg (7,5 mL)
  Interventions: Drug: Nitisinone, suspension

INTERVENTIONS:
Drug: Nitisinone, capsule
  Arms: Orfadin capsules, fasting
Drug: Nitisinone, suspension
  Arms: Orfadin suspension, fasting; Orfadin suspension, with food

SUMMARY:
The study is primarily being performed in order to demonstrate bioequivalence between the Orfadin (nitisinone) suspension and the marketed capsule formulation. The study will also contain a comparison of the bioavailability of the suspension given with food and on an empty stomach.

DETAILED DESCRIPTION:
This is an open, randomized 3-way crossover study in 12 healthy volunteers. Subjects will receive single oral 30-mg doses of nitisinone as a suspension (fasting and with food) and as hard gelatin capsules (fasting only). There will be a 2-week washout period between the doses.

There will be a screening visit within 3 weeks prior to the first dose. During each treatment period, subjects will be admitted to the clinic from the afternoon on the day before drug administration (i.e., on Day -1) and remain at the clinic until the 48-hour post-dose blood sample has been collected in the morning of Day 3. They will then return for ambulatory visit in the morning of Day 4 (72-hour sample). A follow-up visit will take place 7-14 days after the last dose.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers
* Age: 18-55 years, inclusive
* BMI: 18,5-30,0 kg/m2, inclusive

Exclusion Criteria:

* heavy smokers
* Consumption of more than 4 cups of coffee per day.
* History of drug and/or alcohol abuse.
* Positive drug screen or alcohol breath test.
* Positive screens for hepatitis B surface antigen, hepatitis C antibodies and human immunodeficiency virus (HIV) 1-2 antibodies.
* Enrollment in another concurrent clinical study
* Intake of an investigational medicinal product within three months prior to inclusion in this study.
* Donation of more than 50 mL of blood within 60 days prior to drug administration
* Donation of more than 1,5 liters of blood in the 10 months prior to first drug administration.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2012-08; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erik Brouwer, MD, Study Director — Swedish Orphan Biovitrum
Locations (1):
- Pharmaceutical Research Associates Group B.V (PRA), Zuidlaren, Netherlands

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First subject screened: 29 August 2012 Last subject last visit: 25 October 2012.
Groups:
- All Treatment Groups: All participants received all study treatments in a randomized fashion. Subjects were allocated to one of the following treatment sequences (2 subjects to each sequence):
  A B C; B C A; C A B; C B A; A C B; B A C where A=Orfadin capsules, single dose, 30 mg; B=Orfadin suspension, single dose 30 mg, fasting; C=Orfadin suspension, single dose 30 mg, fed
Period: Overall Study
Arm/Group | All Treatment Groups
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: All treatment arms
Arm/Group | Overall Study
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 12
Region of Enrollment [Number; unit: participants]
  Netherlands | 12

OUTCOME MEASURES:

1. Primary Outcome: The Area Under the Serum Concentration Curve (AUC) During 72 Hours After Dose (AUC72h) During Fasting Conditions.
Time Frame: Day 1 predose and at 15, 30, 45 minutes and 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 10, 12, 24, 36, 48 and 72 hours postdose.
Population: Full analysis set was used; subjects with available PK data for at least one of the treatments.
Measure: Geometric Mean (Full Range); unit: uM*h
Groups:
- Orfadin Suspension, Fasting: Orfadin suspension 4 mg/mL, single dose, 30 mg (7,5 mL)
Arm/Group | Orfadin Capsules, Fasting | Orfadin Suspension, Fasting
Number analyzed (Participants) | 12 | 12
uM*h | 403 [315 to 500] | 346 [264 to 456]
Statistical Analysis 1: Comparison: Orfadin Capsules, Fasting vs Orfadin Suspension, Fasting; Test type: Non-Inferiority or Equivalence — Bioequivalence was established if the 90% confidence interval of the ratio was completely within the acceptance range (0.80-1.25); ANOVA; Ratio of geometric means = 0.858, 90% CI 2-sided [0.81 to 0.91]

2. Primary Outcome: The Maximum Serum Concentration (Cmax) During Fasting Conditions.
Time Frame: Day 1 predose and at 15, 30, 45 minutes and 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 10, 12, 24, 36, 48 and 72 hours postdose.
Population: Full analysis set was used; subjects with available PK data for at least one of the treatments.
Measure: Geometric Mean (Full Range); unit: nM
Arm/Group | Orfadin Capsules, Fasting | Orfadin Suspension, Fasting
Number analyzed (Participants) | 12 | 12
nM | 10213 [8030 to 18000] | 9741 [7780 to 20300]
Statistical Analysis 1: Comparison: Orfadin Capsules, Fasting vs Orfadin Suspension, Fasting; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Ratio of geometric means = 0.954, 90% CI 2-sided [0.85 to 1.07]

3. Secondary Outcome: The Area Under the Serum Concentration Curve (AUC) During 72 Hours After Dose (AUC72h)
Description: Measured for the Orfadin suspension treatments arms- both fasting and with food.
Time Frame: Day 1 predose and at 15, 30, 45 minutes and 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 10, 12, 24, 36, 48 and 72 hours postdose.
Population: Full analysis set was used; subjects with available PK data for at least one of the treatments.
Measure: Geometric Mean (Full Range); unit: uM*h
Groups:
- Orfadin Suspension, With Food: Orfadin suspension 4 mg/mL, single dose 30 mg (7,5 mL)
Arm/Group | Orfadin Suspension, Fasting | Orfadin Suspension, With Food
Number analyzed (Participants) | 12 | 11
uM*h | 346 [264 to 456] | 350 [251 to 467]
Statistical Analysis 1: Comparison: Orfadin Suspension, Fasting vs Orfadin Suspension, With Food; Test type: Non-Inferiority or Equivalence — Equivalence (no food effect) was established if the 90% confidence interval of the ratio was completely within the acceptance range (0.80 - 1.25); ANOVA; Ratio of geometric means = 1.013, 90% CI 2-sided [0.96 to 1.07]

4. Secondary Outcome: The Maximum Serum Concentration (Cmax)
Description: Measured for the Orfadin suspension treatment arms- both fasting and with food.
Time Frame: Day 1 predose and at 15, 30, 45 minutes and 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 10, 12, 24, 36, 48 and 72 hours postdose.
Population: Full analysis set was used; subjects with available PK data for at least one of the treatments.
Measure: Geometric Mean (Full Range); unit: nM
Arm/Group | Orfadin Suspension, Fasting | Orfadin Suspension, With Food
Number analyzed (Participants) | 12 | 11
nM | 9741 [7780 to 20300] | 7808 [5300 to 12500]
Statistical Analysis 1: Comparison: Orfadin Suspension, Fasting vs Orfadin Suspension, With Food; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; ANOVA; Ratio of geometric means = 0.802, 90% CI 2-sided [0.71 to 0.90]

5. Secondary Outcome: AUC From Time Zero to Infinity
Description: Measured for the Orfadin capsules and suspension treatments arms - both fasting and with food.
Time Frame: Day 1 predose and at 15, 30, 45 minutes and 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 10, 12, 24, 36, 48 and 72 hours postdose.
Population: Per-protocol set (bioequivalence) was used for fasted treatment groups and per-protocol set (food effect) for fed treatment group (all subjects with available PK data)
Measure: Geometric Mean (Full Range); unit: h*uM
Groups:
- Orfadin Suspension, With Food: Orfadin suspension 4 mg/mL, single dose, 30 mg (7,5 mL)
Arm/Group | Orfadin Capsules, Fasting | Orfadin Suspension, Fasting | Orfadin Suspension, With Food
Number analyzed (Participants) | 12 | 12 | 11
h*uM | 633 [366 to 891] | 559 [454 to 715] | 577 [417 to 858]

6. Secondary Outcome: Time to Reach C-Max (t-Max)
Description: Measured for the Orfadin capsules and suspension treatments arms - both fasting and with food.
Time Frame: Day 1 predose and at 15, 30, 45 minutes and 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 10, 12, 24, 36, 48 and 72 hours postdose.
Population: Per protocol set (bioequivalence) was used for fasting treatments and per protocol set (food effect) used for fed treatment (all subjects with available PK data)
Measure: Median (Full Range); unit: hours
Arm/Group | Orfadin Capsules, Fasting | Orfadin Suspension, Fasting | Orfadin Suspension, With Food
Number analyzed (Participants) | 12 | 12 | 11
hours | 3.50 [0.75 to 8.00] | 0.38 [0.25 to 4.00] | 8.00 [3.50 to 10.00]

7. Secondary Outcome: Terminal Half-life
Description: Measured for the Orfadin capsules and suspension treatments arms - both fasting and with food.
Time Frame: Day 1 predose and at 15, 30, 45 minutes and 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 10, 12, 24, 36, 48 and 72 hours postdose.
Population: as for outcome 6
Measure: Median (Full Range); unit: hours
Groups:
- Orfadin Suspension, Fasting; Orfadin Suspension, With Food: Orfadin suspension 4 mg/mL, single dose, 30 mg (7.5 mL)
Arm/Group | Orfadin Capsules, Fasting | Orfadin Suspension, Fasting | Orfadin Suspension, With Food
Number analyzed (Participants) | 12 | 12 | 11
hours | 48.7 [20.6 to 66.4] | 53.6 [39.3 to 63.7] | 54.3 [37.3 to 75.6]

8. Secondary Outcome: Oral Clearance (CL/F)
Description: Measured for the Orfadin capsules and suspension treatments arms - both fasting and with food.
Time Frame: Day 1 predose and at 15, 30, 45 minutes and 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 10, 12, 24, 36, 48 and 72 hours postdose.
Population: as for outcome 6
Measure: Median (Full Range); unit: L/h
Groups:
- Orfadin Suspension, Fasting: Orfadin suspension, 4 mg/mL, single dose, 30 mg (7.5 mL)
Arm/Group | Orfadin Capsules, Fasting | Orfadin Suspension, Fasting | Orfadin Suspension, With Food
Number analyzed (Participants) | 12 | 12 | 11
L/h | 0.145 [0.102 to 0.249] | 0.160 [0.127 to 0.201] | 0.158 [0.106 to 0.218]

9. Secondary Outcome: Apparent Volume of Distribution (Vz/F)
Description: Measured for the Orfadin capsules and suspension treatments arms - both fasting and with food.
Time Frame: Day 1 predose and at 15, 30, 45 minutes and 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 10, 12, 24, 36, 48 and 72 hours postdose.
Population: as for outcome 6
Measure: Median (Full Range); unit: L
Arm/Group | Orfadin Capsules, Fasting | Orfadin Suspension, Fasting | Orfadin Suspension, With Food
Number analyzed (Participants) | 12 | 12 | 11
L | 9.80 [7.42 to 12.0] | 12.2 [8.59 to 16.7] | 12.8 [8.48 to 17.2]

ADVERSE EVENTS:
Arm/Group | Orfadin Capsules, Fasting | Orfadin Suspension, Fasting | Orfadin Suspension, With Food
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 1/12 | 2/12 | 2/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Orfadin Capsules, Fasting (N=12) | Orfadin Suspension, Fasting (N=12) | Orfadin Suspension, With Food (N=12)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Catheter site related reaction (General disorders) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days